CLINICAL TRIAL: NCT06569069
Title: Effectiveness of Ultrasound-guided Percutaneous Electrolysis Compared to Placebo Acupuncture in Posterolateral Lumbar Disc Herniation: Randomized Controlled Trial
Brief Title: Ultrasound-guided Percutaneous Electrolysis Compared to Placebo Acupuncture in Posterolateral Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Dr. Pablo Herrero Gallego, Physiotherapist, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UG-PE in Disc Herniation
Record Dates: First submitted 2024-08-22; First posted 2024-08-23 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Posterolateral Disc Herniation L4-L5-S1; Disk Herniated Lumbar
Keywords: disc herniation; US guided PE; Lumbar pain
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-guided PE (Experimental)
  Interventions: Other: US guided PE
- Sham acupuncture group (Sham Comparator)
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Other: US guided PE — The multifidus muscle near the posterior dorsal root (at L4-L5 or L5-S1) was targeted using a transverse ultrasound view, inserting the needle at an 80º short axis or a 45º long axis, based on vessel presence. For the tibial nerve in the popliteal region, the needle was inserted at an 80º angle after a transverse cut of the nerve.
  Physio invasiva® needles (0.30 x 40-60 mm) were used in the lumbar region, and 0.30 x 30 mm needles in the popliteal region. Both areas received galvanic current (1.5 mA for three seconds and three impacts). Treatment included three US-guided PE sessions over a 1:7:14 schedule, though two participants skipped the third due to pain resolution.
  Arms: US-guided PE
Other: Sham Acupuncture — Participants in the control group were also treated in a prone position. Sham acupuncture treatment was applied at the superficial level of the posterior face of the thigh on the affected side, using five "Agupunt®" needles of 0.16 x 25 mm, inserted superficially in the lateral aspect of the lumbar area (L3-L4), lateral gluteal region, greater trochanter, lateral part of the distal third of the thigh, head of the fibula and lateral aspect of the leg in its middle third. The needles were left superficially subcutaneously for 15 minutes, performing this approach in three different sessions, again following a periodicity of 1:7:14 days.
  Arms: Sham acupuncture group

SUMMARY:
Lumbar discopathies are among the most common medical concerns in Europe and Spain. Globally, around 2-3% of the population is affected by this condition, which manifests as tingling, burning, itching, muscle weakness, limb pain, or allodynia. The most frequent cases involve lumbar disc herniations at the L4-L5 and L5-S1 levels, which typically compress the tibial nerve. This nerve provides motor and sensory innervation to the posterior knee, leg, foot sole, and posterior thigh.

Treatment options for lumbar discopathies range from pharmacological interventions (cytokine inhibitors, analgesics, muscle relaxants, corticosteroids, non-steroidal anti-inflammatory drugs, and vitamin B12), to ozone injections, nerve root blocks, or surgeries like discectomy. However, conservative physiotherapy approaches, such as therapeutic exercise, axial decompression, transcutaneous electrical nerve stimulation, and peripheral electric stimulation, have gained attention for their efficacy in treating lumbar discopathy symptoms.

Physiotherapy uses electrical currents, applied either directly via needles under ultrasound guidance or non-invasively, to improve the quality of life for individuals with lumbar-origin peripheral nerve involvement. Ultrasound-guided percutaneous electrolysis (US-guided PE) is being explored for its fibrolytic effects in areas of tendon-nerve fibrosis, such as the proximal hamstring tendon and sciatic nerve, and its potential influence on the autonomic nervous system. This suggests that PE might depolarize peripheral nerve synapses, alleviating chronic irritability.

Although Valera et al. have investigated ultrasound-guided PE for neuropathies through the multifidus muscles, no studies have yet focused on PE near the tibial nerve, despite its high incidence in lumbar discopathy cases. Therefore, this study aimed to evaluate the effectiveness of US-guided PE on the tibial nerve in improving pain and muscle strength in patients with L4-L5 or L5-S1 posterolateral disc herniation compared to sham acupuncture.

DETAILED DESCRIPTION:
The study aimed to assess the effectiveness of ultrasound-guided percutaneous electrolysis (US-guided PE) in reducing pain and improving muscle strength in individuals with posterolateral lumbar disc herniations compared to placebo acupuncture.

To achieve this, a randomized, placebo-controlled, single-blindedclinical trial is proposed with two study groups:

* US-guided PE:
* Placebo acupuncture Participants in both groups received 3 sessions with periodicity 1:7:14, meaning seven days elapsed between the first and second sessions, and 14 days between the second and third sessions.

ELIGIBILITY:
Inclusion Criteria:

* positive Lasegue and/or Bragard tests
* presence of posterolateral disc herniation of the L4-L5 and/or L5-S1 vertebral segment of more than 3 months of evolution diagnosed by magnetic resonance imaging
* presence of neuropathic symptomatology in the path of the tibial nerve

Exclusion Criteria:

* belonephobia
* cardiovascular or nervous pathology of medical relevance
* surgical history in the lumbar region
* pregnant women
* recent or current oncologic treatment (for at least 6 months)
* poor echogenicity in the ultrasound image of the areas to be treated

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Low back pain intensity | Measurements will be taken before intervention and four weeks after the third session (last session) of treatment
  This will be measured using the Visual Analogue Scale (minimum score 0, maximum score 10, higher values means worse pain)

SECONDARY OUTCOMES:
Neuropathic symptoms | Measurements will be taken before intervention and four weeks after the third session (last session) of treatment
  This will be measured using the Doleur Neuropatique 4 questionnaire (minimum score 0, maximum score 10, higher values means more neuropathic symtoms)
Hamstrings strength | Measurements will be taken before intervention and four weeks after the third session (last session) of treatment
  This will be measured using the manual muscle testing (minimum score 0, maximum score 5, higher values means more strength).
Triceps suralis strength | Measurements will be taken before intervention and four weeks after the third session (last session) of treatment
  This will be measured using the manual muscle testing (minimum score 0, maximum score 5, higher values means more strength).
Posterior Tibialis strength | Measurements will be taken before intervention and four weeks after the third session (last session) of treatment
  This will be measured using the manual muscle testing (minimum score 0, maximum score 5, higher values means more strength).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Herrero, Study Director — Universidad de Zaragoza
Locations (1):
- University of Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a reasonable request contacting with the main author once data has been published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once research has been published
Access Criteria: Study protocol will be publish in a scientific journal